CLINICAL TRIAL: NCT05528796
Title: Uncovering the Etiologies of Non-immune Hydrops Fetalis Through Comprehensive Genomic Analyses and Phenotyping
Brief Title: Uncovering the Etiologies of Non-immune Hydrops Fetalis
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); University of California, San Diego (Other); Albert Einstein College of Medicine (Other); Johns Hopkins University (Other); University of Pennsylvania (Other); The Jackson Laboratory (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: R01HD107190 (NIH); R01HD107190 (NIH)
Record Dates: First submitted 2022-09-01; First posted 2022-09-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Non-Immune Hydrops Fetalis
MeSH Terms: conditions — Hydrops Fetalis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Pregnancies where the fetus has been diagnosed with NIHF (Experimental): The unit of analysis will be the "proband", i.e. pregnancy/fetus affected with non-immune hydrops fetalis (NIHF).
  Pregnant individuals receiving care at one of the participating sites whose fetus has been diagnosed with NIHF of unknown etiology will be eligible for recruitment and enrollment in this study. Biological fathers of the fetus with NIHF will also be enrolled when available in order to determine inheritance of fetal genetic variants when identified.
  Interventions: Diagnostic Test: Whole genome sequencing

INTERVENTIONS:
Diagnostic Test: Whole genome sequencing — The investigators will study the genes in a fetus' or child's DNA using a test called genome sequencing. Genes are the instructions passed from individuals to a child, and genes determine how bodies are built and grow. Some medical conditions are caused by differences in genes, and the genome sequencing test looks for changes in genes and other parts of a person's genetic sequence (the genome).
  Genetic material will be extracted from bio-specimens. Genome sequencing for this study will be performed at the UCSF Genomic Medicine Laboratory at UCSF. When the genome sequencing results are available, the investigators will arrange an in person or telehealth meeting to explain the test results and what the results mean for the fetus, pregnancy, and family.

SUMMARY:
Non-immune hydrops fetalis (NIHF) is diagnosed on prenatal ultrasound when abnormal fluid collections are seen in the fetus. NIHF carries significant risks of stillbirth, preterm birth, and postnatal morbidity and mortality, particularly when the etiology remains unknown and critical opportunities for focused care and implementation of treatments are missed. In contrast, when an etiology is found, both pre- and postnatal management are directly impacted: counseling is focused, risks to the fetus and neonate are accurately anticipated, surveillance and in utero available treatments such as intrauterine transfusions are implemented, and postnatal treatments are promptly initiated to optimize outcomes. The overarching hypothesis is that discovering the precise etiologies of NIHF will create critical opportunities to improve outcomes through earlier, targeted pre- and postnatal care. Several important steps remain in order to uncover the genetic etiologies for cases remaining unsolved and improve care for these pregnancies. The study team proposes a multicenter collaboration to discover additional genetic diseases and novel variants underlying NIHF in a prospectively enrolled, large and diverse cohort utilizing whole genome sequencing (WGS) and RNA sequencing. The team will further perform comprehensive phenotyping to: a) collect detailed postnatal phenotypes and outcomes, b) re-analyze WGS data utilizing postnatal phenotype to identify diagnoses missed when sequencing algorithms incorporated only phenotype, and c) expand the phenotypes of all genetic in utero in utero diseases the investigators identify to optimize prenatal diagnosis and yield of genomic testing during pregnancy. Such a focused and comprehensive approach to the evaluation and diagnosis of NIHF has not previously been performed, particularly in a large and diverse cohort, and it is expected that this work will significantly improve the ability to understand and reshape the perinatal care for NIHF. This work will lay the foundation for redefining the approach to prenatal diagnosis, management, in utero and postnatal care for NIHF, and will create future opportunities to develop novel diagnostic algorithms and approaches to manage the complications of specific diseases underlying in utero NIHF.

DETAILED DESCRIPTION:
The etiology of non-immune hydrops fetalis (NIHF) remains unknown in at least half of all cases after standard prenatal testing; the comprehensive approach with genomic testing and detailed phenotyping is critical for better understanding this highly morbid condition and ultimately improving outcomes. NIHF occurs in up to 1 in 1700 pregnancies and is diagnosed when abnormal fetal fluid collections (such as pericardial effusion, pleural effusion, ascites, and skin edema) are detected on prenatal ultrasound. Risks include preterm birth in 57-80% of cases, stillbirth in 17-30%, and neonatal death in 29-50%. When the etiology is unknown, critical pre- and postnatal opportunities for focused care and prompt initiation of available treatments are missed. In contrast, when an etiology such as a hereditary anemia or lysosomal storage disorder is found, prenatal counseling is focused, risks to the fetus and neonate are accurately anticipated, in utero surveillance and available treatments such as intrauterine transfusions are implemented, and postnatal treatments are promptly initiated to optimize outcomes.

Many genetic etiologies may underlie NIHF, particularly single gene disorders missed by standard microarray and karyotype. Exome sequencing (ES), whole genome sequencing (WGS), and functional studies are emerging tools for prenatal diagnosis. ES examines >20,000 genes, WGS examines these genes as well as other structural genomic changes, and functional studies such as RNA sequencing evaluate downstream effects of genomic changes. Prior to this work, these approaches had not been used to study NIHF. In a preliminary study of 127 NIHF cases unexplained by standard genetic testing, the study team identified diagnostic variants in 29% with ES and a variant of potential significance in another 9%. This yield is much higher than the 8.5-10% reported for all fetal anomalies with ES, highlighting the burden of single gene disorders in NIHF. The study team identified genetic diseases with greatly variable ultimate severity as well as pre- and postnatal management. However, important steps remain to improve care for these cases: identify additional underlying genetic variants, structural rearrangements, and candidate genes to more fully understand the genetic etiologies of NIHF; enroll a larger, racially diverse cohort to decrease disparities in disease identification; and comprehensively describe in utero and postnatal features of genetic diseases manifesting with NIHF to expand knowledge of their perinatal phenotypes and optimize the yield of prenatal sequencing.

The overarching hypothesis is that discovering the precise etiologies of NIHF will create critical opportunities to improve outcomes through earlier, targeted pre- and postnatal care. The HyDROPS study (Hydrops: Diagnosing and Re-defining Outcomes with Precision Study) where 127 cases were sequenced was conducted by the PI, and the expert multidisciplinary team is ideally positioned to carry the next steps (HyDROPS2) forward. The study will enroll from 5 large medical centers across the country to increase racial and ancestral diversity of the cohort to thoroughly elucidate genetic diseases underlying NIHF, and perform detailed in utero and postnatal phenotyping to improve the accuracy of prenatal diagnosis. The specific aims of the study are:

Specific Aim 1: Discover additional genetic diseases and novel genomic variants underlying NIHF with WGS and RNA sequencing in a large, diverse cohort. Aim 1A) Uncover novel genomic variants with WGS in HyDROPS cases not explained by ES. Aim 1B) Identify novel genomic variants with WGS as well as functional consequences of selected variants with RNA sequencing in a large, prospectively enrolled, racially diverse HyDROPS2 cohort. It is expected to identify a diagnostic variant in 40% of all unexplained NIHF cases with WGS, a diagnostic variant in 10% of cases selected to undergo RNA sequencing, as well as many additional diseases and genomic variants that are critical for understanding the etiologies of NIHF.

Specific Aim 2: Characterize the pre- and postnatal phenotypes for NIHF cases in HyDROPS and HyDROPS2 to expand knowledge of disease-specific features and optimize diagnostic accuracy. Aim 2A) Describe postmortem features for demises and longer term outcomes for living cases to capture phenotypic data missed in utero. Aim 2B) Re-analyze prenatal WGS data using postnatal phenotype to identify diagnoses missed when only the in utero phenotype was incorporated. Aim 2C) Characterize the prenatal phenotypic features for the full spectrum of genetic diseases the investigators diagnose underlying NIHF. It is expected that a substantial proportion of cases will have additional postnatal phenotype important for accurate disease identification, that re-analyzing WGS data utilizing postnatal phenotype will yield a diagnosis in 20% of originally negative or inconclusive cases, and that many in utero features of genetic diseases are underrecognized and thus limit accurate prenatal diagnosis.

Through these aims, the study team will gain a much deeper understanding of the genomic etiologies and disease-specific in utero features of NIHF. This will lay the groundwork to redefine the prenatal approach to NIHF through earlier and accurate diagnosis, and to develop novel, disease-specific in utero management strategies. This precision approach will improve the course for fetuses and families encountering NIHF.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant individuals whose fetus has been diagnosed with NIHF and standard prenatal testing with karyotype and/or microarray is non-diagnostic
* Neonates who received a prenatal diagnosis of NIHF, but genetic testing was unable to be completed or was deferred until after delivery
* Biological parents of the fetus or neonate with NIHF will be enrolled; there are no further inclusion or exclusion criteria for biological parents

Exclusion Criteria:

• Fetuses/neonates with prenatal presentation of

* hydrops secondary to twin-twin transfusion syndrome,
* a clear viral etiology, or
* alloimmunization.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Number of cases for whom a genetic disease or novel variants were identified for underlying NIHF | 1-3 months
  Cases with NIHF for whom pathogenic or likely pathogenic variants were identified implicating genetic disease

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Sparks, MD, Principal Investigator — UCSF Department of Obstetrics, Gynecology and Reproductive Sciences
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No